CLINICAL TRIAL: NCT02319408
Title: A Randomized Phase II Study of Radiation Induced Immune Boost in Operable Non-small Cell Lung Cancer
Brief Title: Immune Boost In Non-Small Cell Lung Cancer
Acronym: RadImmune
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Cancer Research Center (Other); Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. med. Seyer Safi, Dr. med. Seyer Safi, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S-576/ 2013
Record Dates: First submitted 2014-05-27; First posted 2014-12-18 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No radiation (No Intervention): Lobectomy for lung cancer without preoperative radiation
- Preoperative radiation (Experimental): Lobectomy for lung cancer with preoperative radiation
  Interventions: Radiation: Preoperative radiation

INTERVENTIONS:
Radiation: Preoperative radiation — Lobectomy for lung cancer following preoperative radiation
  Arms: Preoperative radiation

SUMMARY:
Insufficient migration and activation of tumour specific effector T cells seems to be the one important reason for inadequate host anti-tumour immune response. Ionizing radiation can induce a variety of immune responses. The goal of this randomized trial is to assess if a preoperative single fraction low dose radiation is able to improve anti-tumour immune response in operable early stage lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven clinical stage I to IIA pulmonary adenocarcinoma
* Lung tumor is felt to be curatively resectable by the treating physicians
* Sufficient pulmonary function for lobectomy according to current guidelines
* The patient is free of distant metastases as confirmed by contrast-enhanced chest and upper abdomen CT-scan and by contrast-enhanced CT or MRI of the brain
* Age over 50years at the time of consent due to federal radiation protection law
* In female patients of childbearing potential there must be a negative pregnancy test
* Eastern Cooperative Oncology Group performance status of 0,1, 2 or 3 at the time of randomization
* Patients who the investigator believes can and will comply with the requirements of this protocol
* Written informed consent according to good clinical practise and national/regional regulations

Exclusion Criteria:

* The patient shows clinical signs of pneumonia
* The patient receives immunosuppressive drugs (alkylating agents, antimetabolites, methotrexate, azathioprine, mercaptopurine, cytotoxic antibodies, ciclosporin, tacrolimus, sirolimus, interferon, mycophenolate, small biological agents)
* The patient has been diagnosed with a potential immune mediated disease
* Elevated blood leukocyte count or erythrocyte sedimentation rate
* Pregnancy
* The patient has received any cancer specific treatment, including radiotherapy, immunotherapy, hormonal therapy or chemotherapy
* The patient is diagnosed with a concomitant malignancy and/or has a history of malignancy within the past five years or has had a malignancy that has been in complete remission for less than 5 years
* The patient needs chronic long term oxygen therapy
* The patient has undergone splenectomy
* The patient is known to be HIV positive
* The patient has an uncontrolled bleeding disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-04; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Cluster of differentiation (CD)8+ T cells in resected NSCLC | 7 days
  Frequencies of CD8+ T cells in resected NSCLC tumors determined by immunohistochemistry

SECONDARY OUTCOMES:
T cell subtypes in resected NSCLC | 7 days
  Frequencies of CD3+, CD4+, CD45RO and Foxp3+ T cells in resected NSCLC tumors determined by immunohistochemistry and flow cytometry

OTHER OUTCOMES:
Tumor reactive T cells | 3 months
  Frequencies of tumor reactive T cells in blood and bone marrow before radiotherapy and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Seyer Safi, MD, PhD, Principal Investigator — University Hospital Heidelberg; Hans Hoffmann, MD, PhD, Principal Investigator — University Hospital Heidelberg; Peter Huber, MD, PhD, Principal Investigator — German Cancer Research Centre
Locations (2):
- Germany (2):
  - Department of Thoracic Surgery, Thoraxklinik, University Hospital Heidelberg, Heidelberg
  - German Cancer Research Centre and Clinic for Radiation Oncology of the University of Heidelberg, Heidelberg

REFERENCES:
- [Background] Klug F, Prakash H, Huber PE, Seibel T, Bender N, Halama N, Pfirschke C, Voss RH, Timke C, Umansky L, Klapproth K, Schakel K, Garbi N, Jager D, Weitz J, Schmitz-Winnenthal H, Hammerling GJ, Beckhove P. Low-dose irradiation programs macrophage differentiation to an iNOS(+)/M1 phenotype that orchestrates effective T cell immunotherapy. Cancer Cell. 2013 Nov 11;24(5):589-602. doi: 10.1016/j.ccr.2013.09.014. Epub 2013 Oct 24. PMID 24209604
- [Result] Safi S, Beckhove P, Warth A, Benner A, Roeder F, Rieken S, Debus J, Dienemann H, Hoffmann H, Huber PE. A randomized phase II study of radiation induced immune boost in operable non-small cell lung cancer (RadImmune trial). BMC Cancer. 2015 Dec 19;15:988. doi: 10.1186/s12885-015-2006-2. PMID 26686362